CLINICAL TRIAL: NCT05482126
Title: Sensory Filtering in the Human Basal Ganglia as a Mechanism of Parkinson's Disease
Status: Recruiting | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Zachary Irwin, Assistant Professor, University of Alabama at Birmingham
Other Study IDs: IRB-300008936; R01NS124563 (NIH)
Record Dates: First submitted 2022-07-26; First posted 2022-08-01 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Parkinson Disease
Keywords: Parkinson; Sensory Processing; Basal Ganglia; Deep Brain Stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Deep Brain Stimulation Surgery Patients: The investigators will seek to enroll people with Parkinson's disease (PD) who have been approved for deep brain stimulation surgery (DBS) as part of their routine clinical
  Interventions: Diagnostic Test: Intraoperative Behavioral Testing; Diagnostic Test: Behavioral Testing
- Healthy controls: The investigators will seek to enroll a cohort of age- and sex-matched healthy individuals to act as a control group. This group will NOT undergo DBS surgery
  Interventions: Diagnostic Test: Behavioral Testing

INTERVENTIONS:
Diagnostic Test: Intraoperative Behavioral Testing — During DBS surgery, tasks will be administered via a tablet PC or mounted monitor, and the subject may hold a response box, joystick, or dynamometer to record responses. During task periods, sensory stimuli will be delivered to the participant, who may be asked to perform a motor behavior in response. Stimuli will consist of audiovisual cues presented on a computer screen, vibration applied to specific parts of the body via a tactor, mild electrical pulses delivered through the skin of specific parts of the body via the attached EMG electrodes, and/or a movement of the arm or joint. Motor responses will consist of simple movements such as finger-tapping or hand-opening, or use of a joystick or dynamometer to move a computer cursor on the screen. Participants may be asked to respond only to a particular sensory stimulus and ignore others, in order to modulate the relevance of each stimulus to the task.
  Groups: Deep Brain Stimulation Surgery Patients
Diagnostic Test: Behavioral Testing — In the lab, tasks will be administered via a tablet PC or mounted monitor, and the subject may hold a response box, joystick, or dynamometer to record responses. During task periods, sensory stimuli will be delivered to the participant, who may be asked to perform a motor behavior in response. Stimuli will consist of audiovisual cues presented on a computer screen, vibration applied to specific parts of the body via a tactor, mild electrical pulses delivered through the skin of specific parts of the body via the attached EMG electrodes, and/or a movement of the arm or joint. Motor responses will consist of simple movements such as finger-tapping or hand-opening, or use of a joystick or dynamometer to move a computer cursor on the screen. Participants may be asked to respond only to a particular sensory stimulus and ignore others, in order to modulate the relevance of each stimulus to the task.

SUMMARY:
The investigators are investigating the brain activity associated with sensory information in movement disorders in order to improve treatment of these symptoms beyond what is currently available.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the functional role of the human basal ganglia in the sensorimotor system. In particular, the investigators are interested in the possibility that the basal ganglia participate in "filtering out" sensory stimuli that are irrelevant to the current behavioral goal. Additionally, the investigators are interested in how this type of sensorimotor processing in these brain areas is related to the severity of movement disorders such as Parkinson's disease and essential tremor.

To do this, the investigators will study both healthy individuals and Parkinson's disease patients undergoing routine deep brain stimulation (DBS) surgery. During the surgery, investigators will place the DBS electrode as routinely performed and additionally place an extra, temporary "strip" electrode along the surface of the brain. Participants will then perform a short behavioral task testing sensorimotor function while investigators record the neural signals from these electrodes. The task will involve the delivery of sensory stimuli (visual, vibrotactile, electrical, and/or proprioceptive), to which the participant will be asked to perform a certain motor response. In order to fully measure the variables of interest, investigators will also attach small stickers (electrodes) to the skin of areas involved in movements for measuring muscle activity (such as the face and limbs), and may attach small, noninvasive devices around the wrist, finger, or arm (e.g., accelerometers) that measure position. The investigators may also apply EEG electrodes to the scalp to measure global brain activity or place a microphone in front of the subject to record speech.

In addition to recording this baseline brain activity, the investigators will evaluate whether deep brain stimulation and dopaminergic medication alters the recorded activity and task performance. Typical deep brain stimulation involves administering specific parameters of high-frequency electrical pulses to achieve clinical benefit. Routine operations involve testing these parameters in the OR in awake patients. For this study, investigators will administer either this high-frequency stimulation or various other patterns of stimulation (e.g., low-frequency, burst stimulation) and measure the changes in behavior and brain activity. As a method of validation, the investigators will also deliver paired pulses of stimulation that enable analysis of stimulation-evoked activity.

Finally, the investigators will correlate recorded brain activity with measures of participants' individual disease severity.

ELIGIBILITY:
Inclusion criteria (PD participants):

1. Age >18 years
2. Clinically definite, advanced idiopathic PD based on consensus criteria.
3. Normal, or essentially normal, preoperative brain MRI.
4. Patient is available for follow-up visits over the length of the study
5. Patient has elected to undergo DBS surgery as part of routine care, and subthalamic nucleus (STN) is determined as the appropriate surgical target

Inclusion criteria (control participants):

1. Age >18 years.
2. No diagnosis of PD, other movement disorder, or other significant neurological disease.

Exclusion criteria (PD participants):

1. Age <18 years.
2. Medical contraindications such as current uncontrolled hypertension, heart disease, coagulopathy, or other conditions that might increase the risk of surgery
3. Diagnosis or suspicion of atypical Parkinsonism (PSP, MSA, CBD) or drug-induced Parkinsonism, or significant neurological disease other than PD.
4. Diagnosis of psychogenic movement disorder based on consensus criteria
5. Prior DBS surgery or ablation
6. Clinical dementia and/or Dementia Rating Scale (DRS) score of <5th percentile adjusted for age and education level, based upon routine pre-op NP testing.
7. Unable to withhold dopaminergic medications for at least 12 hours prior to scheduled visit

Exclusion criteria (control participants):

1. Age <18 years.
2. Previous diagnosis of PD, other movement disorder, or other significant neurological disease.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's disease (PD) who have been approved for deep brain stimulation surgery (DBS) as part of their routine clinical care, as well as healthy controls with no known movement disorder diagnoses
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-06-08 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Kinematic response to stimulus (intraoperative) | Intraoperative
  Arm movements (hand position, velocity) recorded following stimulus onset, measured by joystick outputs.
Kinematic response to stimulus (postoperative) | 1 month post-op
  Arm movements (hand position, velocity) recorded following stimulus onset, measured by joystick outputs.
Latency of response to stimulus (intraoperative) | Intraoperative
  Time from stimulus onset to start of motor response, measured by electromyography (EMG)
Latency of response to stimulus (postoperative) | 1 month post-op
  Time from stimulus onset to start of motor response, measured by electromyography (EMG)
Neural response to stimulus | Intraoperative
  Brain activity recorded following stimulus onset, measured by local field potentials recorded from the electrocorticography (ECoG) and DBS electrodes.

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Irwin, PhD, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- The University of Alabama at Birmingham Hospital, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No